CLINICAL TRIAL: NCT06052670
Title: Functional Diagnostic Accuracy of Ultrasonic Flow Ratio in Assessment of De Novo Coronary Artery Lesions
Brief Title: Functional Diagnostic Accuracy of Ultrasonic Flow Ratio in Assessment of Coronary Artery Lesions
Acronym: FUNCTION
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-GSP-GG-4
Record Dates: First submitted 2023-09-12; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Stenosis
Keywords: intravascular ultrasound; ultrasonic flow ratio; fractional flow reserve
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: fractional flow reserve (FFR); ultrasonic flow ratio (UFR); intravascular ultrasound (IVUS) — pressure wire-based fractional flow reserve (FFR); intravascular ultrasound (IVUS)-based ultrasonic flow ratio (UFR)

SUMMARY:
This is a prospective, single-center study. The primary purpose of this study is to evaluate the sensitivity and specificity of offline computational ultrasonic flow ratio (UFR) with conventional pressure wire-based fractional flow reserve (FFR) as the standard reference. The study will be conducted in Fuwai Hospital, and a total of 408 patients with coronary vessel diameter stenosis ≥30% and ≤80% are planned to be recruited. Participants who meet the inclusion criteria and do not meet the exclusion criteria will undergo intravascular ultrasound (IVUS) followed by FFR examination. IVUS imaging will be sent to an independent core laboratory for UFR calculation. UFR analyses were performed offline in a blinded fashion without awareness of FFR measurement. Using FFR≤0.80 as the gold standard, the sensitivity and specificity of UFR in the functional significance of coronary artery stenosis will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina pectoris, unstable angina pectoris, or after the acute phase of myocardial infarction
* Age ≥18 years
* Written informed consent
* Intermediated coronary lesions (diameter stenosis of 30%-80% by visual estimation from coronary angiography)

Exclusion Criteria:

* Ineligible for diagnostic IVUS or FFR examination
* Prior coronary artery bypass grafting of the interrogated vessels
* Myocardial infarction within 72 h of coronary angiography
* Severe heart failure
* Serum creatinine levels >150 umol/L, or glomerular filtration rates <45 ml/kg/1.73 m2
* Allergy to the contrast agent or adenosine
* Life expectancy < 2 years
* IVUS pullback not covering the entire lesion
* Severe myocardial bridge in the interrogated vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years of age who will be admitted for coronary angiography and had an indication for FFR measurement at the FuWai Hospital, Beijing, China, due to stable angina or unstable angina will be consecutively enrolled.
Sampling Method: Probability Sample
Enrollment: 408 (Estimated)
Dates: Start 2023-09-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of UFR in predicting functionally significant coronary stenosis at the patient level, using FFR as the reference standard | Immediately after the procedure
  Sensitivity is defined as the proportion of UFR ≤ 0.80 in patients with hemodynamically-significant stenosis as measured by FFR (FFR ≤ 0.80); specificity is defined as the proportion of UFR > 0.80 in patients without hemodynamically-significant stenosis as measured by FFR (FFR > 0.80).

SECONDARY OUTCOMES:
Sensitivity and specificity of UFR in predicting functionally significant coronary stenosis at the vessel level, using FFR as the reference standard | Immediately after the procedure
  Sensitivity is defined as the proportion of UFR ≤ 0.80 in vessels with hemodynamically-significant stenosis as measured by FFR (FFR ≤ 0.80); specificity is defined as the proportion of UFR > 0.80 in vessels without hemodynamically-significant stenosis as measured by FFR (FFR > 0.8).
Diagnostic accuracy of UFR in predicting functionally significant coronary stenosis at the patient level, using FFR as the reference standard | Immediately after the procedure
  Diagnostic accuracy is defined as UFFR (≤0.80 or >0.80) to identify hemodynamically-significant coronary stenosis with FFR (≤0.8 or >0.8) as the reference standard.
The AUC of UFR for coronary stenosis with FFR as the gold standard | Immediately after the procedure
  AUC is defined as the area under the receiver-operating characteristic curve